CLINICAL TRIAL: NCT07210905
Title: Implementation of the 3-steps Assess-Advise-Refer Exercise (FitARise) Protocol as a Standard Practice in Cancer Care: A Stepped-wedge Cluster Randomized Trial
Brief Title: Implementation of the 3-steps Assess-Advise-Refer Exercise (FitARise) Protocol as a Standard Practice in Cancer Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: UW 24-572
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-02

CONDITIONS: Exercise; Cancer
Keywords: Implementation study; Weight management; Cancer survivorship
MeSH Terms: conditions — Motor Activity; Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will use a stepped wedge cluster randomized controlled trial design in which the intervention is introduced stepwise across study units . After obtaining the consent form from the 9 oncology units, they will be randomized to one of the three roll-out schedules with a 4-month duration each. All the study units will start the trial in a control condition (i.e., no implementation strategies used). At each time point, a new group of 3 study units will cross over from the control condition to the implementation condition, until all sites are receiving the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation condition (Experimental): Under implementation conditions, the FitARise protocol will be implemented in routine oncological clinics using 4 implementation strategies, including audit, feedback, facilitation, and adaptable workflow at the beginning of the study.
  Interventions: Behavioral: 3-step Assess-Advice-Refer
- Control condition (No Intervention): In the control condition, the clinical outpatient operation is performed as usual. The screening tool and referral forms will be provided to the study sites and clinicians are encouraged eligible patients to adopt the FitARise program. Patients referred to JCICC will be managed following the predefined clinical pathway triage system. A briefing session about the purpose of the implementation program and the introduction of the FitARise protocol will be given to the staff at each study unit before the start of the first 4-months control condition. The briefing session will be recorded for the purpose of fidelity assessment.

INTERVENTIONS:
Behavioral: 3-step Assess-Advice-Refer — Four implementation strategies will be conducted individually for each of the study unit at the timepoint when the study unit is being randomly allocated to the implementation condition. For each study unit, all site facilitators will first receive a half-day training. Each study unit under the implementation condition will receive weekly audit and feedback reports to summarize the proportion of eligible patients, proportion of eligible patients being screened, proportion of patients appropriately referred to JCICC. The senior research assistant with a nursing background will receive training and mentoring from the PI and will be the guided facilitator. The guided facilitator will conduct weekly site visits to address operational issues arise during the implementation. Lastly, while the FitARise protocol is standardized and cannot be modified, the routine workflow for each study unit can be adjusted according to its context and resources.
  Other Names: FitARise
  Arms: Implementation condition

SUMMARY:
This study proposes to evaluate the process and outcome of an implementation program designed to implement the American College of Sports Medicine (ACMS)-recommended exercise assessment, advice, and referral instruction as standard practices in routine cancer care.

DETAILED DESCRIPTION:
This study aims to test whether using implementing strategies (audit, feedback, facilitation, and adaptable workflow) to adopt the systematic FitARise protocol increases the proportion of eligible patients assessed, advised, and referred compared to control with the availability of the protocol, but without implementation strategies. This study hypothesizes that implementing strategies to promote the protocol's adoption will increase the proportion of eligible patients assessed and advised by oncologists and the proportion of patients referred to the JCICC exercise-based weight management program. For process evaluation, this study aims to use qualitative methods to assess the experience and response to the implementation program. The primary outcome (the reach measurement) is the percentage of eligible patients assessed, advised, and referred based on predefined BMI scores.

ELIGIBILITY:
Inclusion Criteria (Cancer patients):

* All cancer patients with BMI score>=23;
* Have completed cancer treatment within the past five years;
* At least 18 years old;
* Are literate in Chinese or English;
* Are eligible to attend the intervention program.

Exclusion Criteria (Cancer patients):

* Patients who have completed cancer treatments for more than five years;
* Non-Cantonese, non-Mandarin, non-English speakers.

Inclusion Criteria (Clinical staff):

- All clinical, medical or surgical oncologists at the study units during the study period.

Exclusion Criteria (Clinical staff):

- No exclusion criterial for staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-02-02 (Estimated); Study Completion 2028-02-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of eligible patients | Pre- and post-implementation phase, up to 24 months
  The primary outcome (the reach measurement) is the percentage of eligible patients assessed, advised, and referred based on predefined BMI scores.

SECONDARY OUTCOMES:
Change in referral uptake | Pre- and post-implementation phase, up to 24 months
  The secondary outcome is the uptake of the referral, i.e. the proportion of referred patients accepting the enrolment of the JCICC weight management program. This study also will examine the attendance rates of those enrolled in the weight management program.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Lam, PhD, Principal Investigator — The University of Hong Kong
Locations (8):
- Hong Kong (8):
  - KWH Department of Surgery, Hong Kong
  - PMH Department of Oncology, Hong Kong
  - PYEH Department of Clinical Oncology, Hong Kong
  - QMH Department of Clinical Oncology, Hong Kong
  - QMH Department of Obstetrics and Gynaecology, Hong Kong
  - QMH Department of Surgery, Hong Kong
  - TMH Department of clinical oncology, Hong Kong
  - YCH Surgery Department, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.